CLINICAL TRIAL: NCT03363399
Title: Flow Cytometric Analysis of Peripheral Blood Neutrophil Myeloperoxidase Expression for Ruling Out Myelodysplastic Syndromes: A Pilot Diagnostic Accuracy Study
Brief Title: Flow Cytometric Analysis of Peripheral Blood Neutrophil Myeloperoxidase Expression and Myelodysplastic Syndromes
Acronym: MPO-MDS-PILOT
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC17.249; 2017-A02361-52 (Other: ID RCB)
Record Dates: First submitted 2017-11-17; First posted 2017-12-06 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia
Keywords: Diagnostic accuracy study; Flow cytometry analysis; Myeloperoxidase; Peripheral blood sample
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Flow cytometry analysis of neutrophil myeloperoxidase expression — Flow cytometry analysis of neutrophil myeloperoxidase expression in peripheral blood samples will be performed within 24 h of MDS diagnostic evaluation and blinded to the reference standard. Peripheral blood samples will be collected in 5 ml (EDTA) anticoagulant plastic tubes and processed within 24 h maximum of collection. The samples will be stored at 4°C overnight.
  Blood samples containing at least 105 neutrophils will be incubated with a panel of antibodies conjugated to fluorochromes, according to the manufacturers' recommendations.
  At least 10,000 cell events will be acquired on a 3-laser, 8-color flow cytometer and analyzed using Becton Dickinson (BD) Fluorescence-activated cell sorting (FACS) Diva Software version 6. Each marker will be expressed as median, geometric and arithmetic mean, regular and robust coefficient of variation.

SUMMARY:
Myelodysplastic syndromes (MDS) constitute a heterogeneous group of clonal bone marrow neoplasms that predominate in the elderly, with a median age at diagnosis of 70 years. MDS are characterized by peripheral blood cytopenia and morphologic dysplasia for one or more hematopoietic cell lineage, reflecting ineffective hematopoiesis.

The diagnostic work-up of MDS includes a bone marrow aspirate and biopsy, which is an invasive procedure, for cytomorphologic and cytogenetic evaluations. Because the prevalence of disease is lower than 20% in subjects referred for suspected MDS, many patients are exposed to unnecessary bone marrow aspiration-related discomfort and harms.

An objective assay is highly desirable for accurately ruling out MDS based on peripheral blood samples, which may obviate the need for invasive bone marrow aspiration and biopsy in patients with negative results.

Few studies have investigated the value of peripheral blood flow cytometric analysis for the diagnosis of MDS and/or chronic myelomonocytic leukemia (CMML). Although promising, these studies lacked replication of their results, used a case-control design, which was prone to spectrum bias, or yielded imprecise diagnostic accuracy estimates due to relatively limited sample sizes.

Anecdotal evidence supports the potential of flow cytometric analysis of peripheral blood neutrophil myeloperoxidase expression for the diagnosis of MDS and CMML. Myeloperoxidase is an enzyme synthetized during myeloid differentiation that constitutes the major component of neutrophil azurophilic granules. Myeloperoxidase expression may reflect neutrophil hypogranulation, which is a classical although subjective dysplastic feature of MDS. Flow cytometric analysis of myeloperoxidase expression in bone marrow neutrophil granulocytes has been used for discriminating low versus high grade MDS. Yet a study reporting on the accuracy of flow cytometric analysis of peripheral blood neutrophil myeloperoxidase expression for the diagnosis of MDS is still lacking, to our knowledge.

In this study, the investigators hypothesize that flow cytometric analysis of neutrophil myeloperoxidase expression in peripheral blood may accurately rule out MDS and obviate the need for bone marrow aspiration and biopsy, with sensitivity approaching 100%, in routine practice.

In this observational diagnostic accuracy study, burden will be null for recruited patients. No specific intervention is assigned to participants. All diagnostic testing, procedures, and medication ordering are performed at the discretion of attending physicians. Flow cytometry analysis of peripheral blood neutrophil myeloperoxidase expression will not require additional blood sample. A test result will have no impact on patient management. No follow-up visits are planned in this cross-sectional study.

DETAILED DESCRIPTION:
The primary objective of MPO-MDS-pilot study is to estimate the accuracy of flow cytometric analysis of neutrophil myeloperoxidase expression in peripheral blood for the diagnosis of myelodysplastic syndromes (MDS) and/or chronic myelomonocytic leukemia (CMML).

The secondary objectives are:

1. to provide accuracy estimates for prespecified thresholds of neutrophil myeloperoxidase expression in peripheral blood in ruling out MDS and/or CMML.
2. to estimate the prevalence of alternate diagnosis established by bone marrow cytomorphology.

The MPO-MDS-pilot project is a multicenter, phase II, cross-sectional, diagnostic accuracy study of consecutive unselected patients referred for suspected MDS or CMML.

Screening: All consecutive patients referred to the immuno-hematology lab at the study sites for suspicion of MDS will be screened for eligibility. A lab physician will review inclusion and exclusion criteria, using computerized medical and laboratory records.

Recruitment: Participants will be included in the study once all the screening activities have been conducted and only if the patient meets all inclusion and none exclusion criteria. The consent for flow cytometry analysis of peripheral blood sample and data collection through chart review will be sought under a regime of "non-opposition" (opt-out): after appropriate written information is delivered, cross-sectional data will be collected except in case of opposition from the patient. All patients included in the study will be assigned a unique patient identification number. This number will be used to identify the patient throughout the study.

Index test: Flow cytometry analysis of neutrophil myeloperoxidase expression in peripheral blood will be performed within 24 h of MDS diagnostic evaluation and blinded to the reference standard.

Reference standard: The diagnosis of MDS will be established according to the World Health Organization (WHO) classification, based on clinical data, peripheral blood cytopenia, cytomorphology of peripheral blood and bone marrow aspirate, and cytogenetic analysis. The criteria for MDS diagnosis are 1) the presence of ≥10% dysplastic cells in any hematopoietic lineage, 2) the exclusion of acute myeloid leukemia (defined by the presence of ≥20% peripheral blood or bone marrow blasts), and 3) the exclusion of reactive etiologies of dysplasia. Cytopenia is defined by hemoglobin concentration <10 g/dL, platelet count <100x109/L, and/or absolute neutrophil count <1.8 x109/L. Yet a diagnosis of MDS could be made with milder levels of cytopenia. Idiopathic cytopenia of uncertain significance (ICUS) is defined by unexplained mild persistent cytopenia for at least 6 months and the failure to establish the diagnosis to MDS according to published guidelines. Consistent with WHO classification, MDS subcategorization will rely on the degree of dysplasia (unilineage versus multilineage), blast percentages, presence of ring sideroblasts, and cytogenetic analysis (del(5q)). The criteria for CMML diagnosis are 1) the presence of persistent peripheral blood monocytosis ≥1 x109/L, and 2) monocyte accounting for more than 10% of the white blood cell differential count. Evaluation of bone marrow cytomorphology will be performed prospectively by experienced hematopathologists who are blinded to the index test results.

Patients with confirmed suspicion of MDS: Participants for whom the diagnosis of MDS (or CMML) is confirmed by the reference standard will be categorized as patients with confirmed suspicion of MDS.

Patients with unconfirmed suspicion of MDS: Participants for whom the diagnosis of MDS (or CMML) is ruled out by the reference standard will be categorized as patients with unconfirmed suspicion of MDS. This latter subgroup will include patients with ICUS, as defined in accordance with published guidelines

Follow-up: No follow-up visit is planned in this cross-sectional diagnostic accuracy study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥50 years;
* Clinical suspicion of myelodysplastic syndromes (MDS) and / or chronic myelomonocytic leukemia (CMML);
* Peripheral blood cytopenia defined by hemoglobin concentration <10 g/dL, platelet count <100 x109/L, and/or absolute neutrophil count <1.8 x109/L.

Exclusion Criteria:

* History of or active documented MDS or CMML;
* Admission to the intensive care unit;
* Suspicion of hematological disease other than MDS requiring bone marrow aspirate and/or biopsy (i.e., acute leukemia,…);
* Absolute neutrophil count <0.5 x109/L;
* Not affiliated with a social security system;
* Homelessness;
* Incarcerated;
* Inability to understand research information and/or to provide non-opposition, because of language restriction, dementia, or altered mental status;
* Refusal to participate;
* Previous enrollment in the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants are consecutive unselected adults of 50 years of age or more and who are referred for suspected MDS or CMML. Suspicion of MDS or CMML is based on medical history and peripheral blood cytopenia.
  To be eligible, patients will be required to meet all three inclusion criteria and none of the exclusion criteria. Yet, patients with milder levels of cytopenia might by eligible based on medical history.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2018-09-06 (Actual)

PRIMARY OUTCOMES:
Area under the Receiver Operating Characteristic (ROC) curve of neutrophil myeloperoxidase expression in peripheral blood | Baseline
  The primary outcome is the discrimination of the index test (i.e., flow cytometry analysis of neutrophil myeloperoxidase expression in peripheral blood) for the diagnosis of myelodysplastic syndromes (MDS) or chronic myelomonocytic leukemia (CMLL) quantified by the area under the ROC curve point estimate along with its 95% confidence interval.

SECONDARY OUTCOMES:
Sensitivity point estimates (along with 95% confidence interval) of neutrophil myeloperoxidase expression in peripheral blood for the diagnosis of MDS or CMML | Baseline
Specificity point estimates (along with 95% confidence interval) of neutrophil myeloperoxidase expression in peripheral blood for the diagnosis of MDS or CMML | Baseline
Negative predictive value point estimates (along with 95% confidence interval) of neutrophil myeloperoxidase expression in peripheral blood for the diagnosis of MDS or CMML | Baseline
Positive predictive value point estimates (along with 95% confidence interval) of neutrophil myeloperoxidase expression in peripheral blood for the diagnosis of MDS or CMML | Baseline
Prevalence point estimate (along with 95% confidence interval) for alternate diagnosis established by bone marrow cytomorphology. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Raskovalova, MD, Study Chair — Centre Hospitalier Universitaire Grenoble Alpes, France; Richard Veyrat-Masson, MD, Principal Investigator — Centre Hospitalier Universitaire Clermont-Ferrand, France; Sophie Park, MD, Principal Investigator — Centre Hospitalier Universitaire Grenoble Alpes, France; Marc Berger, MD, Principal Investigator — Centre Hospitalier Universitaire Clermont-Ferrand, France; Jean-Yves Cesbron, MD, Principal Investigator — Centre Hospitalier Universitaire Grenoble Alpes, France; Marie-Christine Jacob, MD, Principal Investigator — Centre Hospitalier Universitaire Grenoble Alpes, France
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire Estaing, Clermont-Ferrand
  - Centre Hospitalier Universitaire Grenoble Alpes, Grenoble

IPD SHARING:
Plan to Share IPD: Yes
The principal investigators will respond directly to data requests by providing a de-identified data set. Individual participant data that underlie the results reported in the published articles (i.e., main text, tables, figures, and appendices) will be supplied.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 12 months after publication of the main findings of the final dataset.
  No end date.
Access Criteria: De-identified data will be available for individual participant data meta-analysis purpose.
  Researchers should submit a methodologically sound proposal that complies with the Preferred Reporting Items for Systematic Review and Meta-Analysis Protocols (PRISMA-P) 2015 statement. Proposals should be directed to TRaskovalova@chu-grenoble.fr. Data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Raskovalova T, Scheffen L, Jacob MC, Vettier C, Bulabois B, Szymanski G, Chevalier S, Gonnet N, Park S, Labarere J. Comparative diagnostic accuracy between simplified and original flow cytometric gating strategies for peripheral blood neutrophil myeloperoxidase expression in ruling out myelodysplastic syndromes. PLoS One. 2022 Nov 18;17(11):e0276095. doi: 10.1371/journal.pone.0276095. eCollection 2022. PMID 36399441
- [Derived] Raskovalova T, Jacob MC, Bulabois CE, Mariette C, Scheffen L, Park S, Labarere J. Flow cytometric analysis of peripheral blood neutrophil myeloperoxidase expression for ruling out myelodysplastic syndromes: a prospective validation study. Ann Hematol. 2021 May;100(5):1149-1158. doi: 10.1007/s00277-021-04446-7. Epub 2021 Feb 10. PMID 33569703